CLINICAL TRIAL: NCT07078799
Title: A Prospective Randomized Comparison of Wavefront-guided LASIK Surgery to Ray Tracing-Guided LASIK Surgery
Brief Title: Wavefront-guided LASIK Surgery Compared to Ray Tracing-Guided LASIK Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Edward E. Manche, Professor of Ophthalmology, Stanford University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81344
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Myopia; Astigmatism
Keywords: Ray tracing-guided LASIK; Wavefront-guided LASIK
MeSH Terms: conditions — Myopia; Astigmatism | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, contralateral fellow eye study comparing ray-tracing guided LASIK in one eye to wavefront-guided LASIK in the fellow eye of participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wavefront-guided laser ablation (Active Comparator): Wavefront-guided LASIK
  Interventions: Procedure: LASIK
- Ray tracing-guided LASIK (Active Comparator): Ray-tracing guided LASIK is being performed in one eye and Wavefront-guided LASIK is being performed in the fellow eye
  Interventions: Procedure: LASIK

INTERVENTIONS:
Procedure: LASIK — Wavefront-guided LASIK is being performed in one eye and Ray-tracing guided LASIK is being performed in the fellow eye
  Arms: Ray tracing-guided LASIK
Procedure: LASIK — Ray-tracing guided LASIK is being performed in one eye and Wavefront-guided LASIK is being performed in the fellow eye.
  Arms: Wavefront-guided laser ablation

SUMMARY:
We are enrolling participants aged 22 and older to have LASIK surgery in both eyes. We will perform wavefront-guided LASIK in one eye and ray tracing-guided LASIK in the fellow eye of each participant. We are trying to see if there are any differences in the efficacy between the two types of LASIK procedures.

DETAILED DESCRIPTION:
We are comparing the outcomes of wavefront-guided LASIK (laser in-situ keratomileusis) and ray tracing-guided LASIK for nearsightedness with and without astigmatism.

Wavefront aberrometry (a non-contact laser measuring device) is an automated device that measures the refractive status of the eye. This data is then transferred to the laser system and calculates a unique treatment to reduce or eliminate your nearsightedness with and without astigmatism (a non-spherical shape).

One eye will be treated with ray tracing-guided LASIK and the other eye treated with the wavefront-guided LASIK. Each participant will receive both wavefront-guided LASIK and ray-tracing guided LASIK. Both wavefront-guided LASIK and ray tracing-guided LASIK are FDA-approved procedures. Both procedures are being performed according to the FDA-approved labeling.

We plan to enroll up to 70 near-sighted study participants to undergo treatment in this clinical research trial.

The choice of which eye receives ray tracing-guided LASIK surgery and which eye receives wavefront-guided LASIK will be randomized (assigned at random) prior to enrollment.

Participants scheduled to undergo LASIK for the correction of myopia (nearsightedness) will be screened for eligibility. Eligible participants will be examined preoperatively to establish a baseline for ocular condition (the general health and glasses prescription of the eyes). Postoperatively, participants will undergo an ophthalmic evaluation (complete eye examination) at regular intervals as specified in this protocol. Re-treatments (a second operation on the same eye for residual nearsightedness, farsightedness and/or astigmatism) will not be allowed during the first twelve months of this study.. If a participant elects to undergo a re-treatment of the initial LASIK surgery prior to the 12-month post-operative visit, the data after the retreatment procedure will be excluded from the study analysis.

The primary aim of the research is to compare outcomes between the two procedures. All of the procedures performed during the study are considered standard of care for LASIK surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22 and older
2. People with healthy eyes:

   1. No abnormal corneal shape
   2. No excessively thin corneas
   3. No eye diseases such as glaucoma or cataracts
3. Nearsightedness between -1.00 diopters and -10.00 diopters.
4. Subjects with less than or equal to 3.00 diopters of astigmatism.
5. Subjects must have similar levels of nearsightedness in each eye.

Exclusion Criteria:

1. Subjects under the age of 22.
2. Subjects with excessively thin corneas.
3. Subjects with topographic evidence of keratoconus.
4. Subjects with ectactic eye disorders.
5. Subjects with autoimmune diseases.
6. Subjects who are pregnant or nursing at the time of surgery. (The FDA-approved labelling indications for LASIK specifically excludes patients who are pregnant or nursing. There is no strict prohibition not to become pregnant during the one year study period)
7. They can not be more than 1.5 diopter of difference between eyes.
8. Subjects with more than 3.00 diopters of astigmatism
9. Subjects with disimilar levels of astigmatism in each eye (They can not have more than 0.75 diopters of difference between eyes) -

Ages: 22 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Uncorrected visual acuity | One year
  Uncorrected visual acuity using ETDRS charts

SECONDARY OUTCOMES:
5 and 25% best corrected low contrast visual acuity | 12 months
  Measurement of the change in 5 and 25% best corrected low contrast visual acuity using ETDRS charts
Achieved versus attempted ablation depth measured by anterior segment OCT | One, three and twelve months
  Measurement of achieved ablation depth by comparing preoperative anterior segment OCT to postoperative anterior segment OCT
Self reported quality of vision and quality of life measures | Three, six and twelve months
  A validated questionnaire will be administered preoperatively and at postoperative months 3, 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Edward E Manche, MD, Principal Investigator — Stanford University
Locations (1):
- Byers Eye Institute at Stanford University School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided